CLINICAL TRIAL: NCT06530771
Title: Multimodality US Based on Angio Planewave Ultrasensitive Imaging and Shear Wave Elastography to Guide the Fine-Needle Aspiration Management of Thyroid Lesions: Focus on the Innovative Microvascular Classification
Brief Title: Multimodality US Based on Angio Planewave Ultrasensitive Imaging and Shear Wave Elastography to Evaluate the Malignancy Risk Value of Thyroid Nodules
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: ZDWY.CSK.008
Record Dates: First submitted 2024-07-29; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2023-12

CONDITIONS: Multimoda Lultasound; Thyroid Cancer; Microvascular Classification
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Malignant thyroid nodules
  Interventions: Diagnostic Test: ultrasound
- Benign thyroid nodules
  Interventions: Diagnostic Test: ultrasound

INTERVENTIONS:
Diagnostic Test: ultrasound — Conventional US, SWE, and AP of thyroid nodules were conducted successively with a Supersonic Aixplorer system (SuperSonic Imagine, Aix-en-Provence, France) using a 5-14 MHz linear transducer.

SUMMARY:
The goal of this clinical trial is to explore the value of a multimodal ultrasound model based on Angio Planewave Ultrasensitive Imaging, Shear Wave Elastography and grayscale ultrasound in the differential diagnosis of benign and malignant thyroid nodules. The main questions it aims to answer are:

Can an innovative ultra-microvascular classification system based on Angio Planewave Ultrasensitive Imaging distinguish between benign and malignant thyroid nodules? How about the performance of multimodal ultrasound model to Guide the Fine-Needle Aspiration Management of Thyroid Lesions?

Participants will:

Undergo grayscale ultrasound, SWE, and Angio Planewave Ultrasensitive Imaging multimodal thyroid ultrasound examination within one week before surgery Undergo surgery and obtain the postoperative pathological diagnosis

ELIGIBILITY:
Inclusion Criteria:

1. age more than 18 years;
2. Voluntarily signed informed consent;
3. Have 1 or more thyroid nodules detectable by ultrasound;
4. participant underwent surgical procedure to confirm the pathologic results

Exclusion Criteria:

1. Nodules are accompanied by large calcifications followed by acoustic shadows
2. History of previous neck surgery or cancer, thyroid medications, radiation or surgical treatment;
3. Poor quality of retained images or non-standard operations (such as intermittent scanning and improper probe compression), and incomplete pathological results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population data for this prospective single-center cohort study were gathered at the Fifth Affiliated Hospital of Sun Yat-sen University.
Sampling Method: Probability Sample
Enrollment: 720 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficacy | one week
  the area under the receiver operating characteristic (ROC) curve (AUC)
Diagnostic efficacy | one week
  sensitivity, specificity, accuracy
positive predictive value (PPV), and negative predictive value (NPV) | one week
  Diagnostic efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Affiliated Hospital Sun Yat-Sen University, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided